CLINICAL TRIAL: NCT01085773
Title: Effects of Nordic Walking and Exercise on Prescription on Glucose Metabolism in Type 2 Diabetes Mellitus: A Randomized Controlled Trial
Brief Title: Effects of Nordic Walking and Exercise on Glucose Metabolism in Type 2 Diabetes Mellitus: A Randomized Controlled Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Collaborators: University of Southern Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2628-04
Record Dates: First submitted 2010-03-11; First posted 2010-03-12 (Estimated); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Type 2 Diabetes; Exercise
Keywords: HbA1c; Type 2 Diabetes; Lifestyle changes; Exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity | interventions — Nordic Walking

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard written information on exercise (No Intervention): The Control group got the diabetes outpatients clinics standard written information on exercise as a part of the treatment for Type 2 Diabetes and were, like other Type 2 Diabetes patients in the clinic, advised at inclusion to be physically active.
- Exercise on Prescription (Experimental): In Denmark, Exercise on Prescription have focused on individual behavioral change and an exercise program for 16 weeks. The physical training consisted of both aerobic and strength training and took place in supervised groups
  Interventions: Behavioral: Exercise on Prescription
- Nordic Walking (Experimental): Nordic Walking is a fitness type of walking; incorporating the use of specially designed walking sticks. Nordic Walking focuses on aerobic training where the additional activity of the arms increases a person's oxygen uptake and energy expenditure.
  Interventions: Behavioral: Nordic Walking

INTERVENTIONS:
Behavioral: Exercise on Prescription — The physical training consisted of both aerobic and strength training and took place in supervised groups.
  Arms: Exercise on Prescription
Behavioral: Nordic Walking — Nordic Walking is a fitness type of walking; incorporating the use of specially designed walking sticks. Nordic Walking focuses on aerobic training where the additional activity of the arms increases a person's oxygen uptake and energy expenditure.
  Arms: Nordic Walking

SUMMARY:
The objective of this randomized controlled trial was to evaluate the effects of two different physical exercise programs aimed at long-term lifestyle changes in physical activity in patients with Type 2 Diabetes, with glucose metabolism evaluated by HbA1c as the primary outcome.

DETAILED DESCRIPTION:
Physical training and exercise is considered a cornerstone in the treatment of Type 2 Diabetes Mellitus.

Programs which include physical activity as a component in the treatment of Type 2 Diabetes as well as other chronic diseases have in Denmark and other countries been based on "Exercise on Prescription schemes". In Denmark, these schemes have focused on individual behavioral change and an exercise program for 16 weeks. No studies have documented whether "Exercise on Prescription" helps patients with Type 2 Diabetes to change their lifestyle behavior or whether it has a positive impact on measurements for physical capacity and glucose metabolism.

Nordic Walking is a fitness type of walking; incorporating the use of specially designed walking sticks. Nordic Walking focuses on aerobic training where the additional activity of the arms increases a person's oxygen uptake and energy expenditure.

In Denmark, many activity programs and concepts such as Exercise on Prescription and Nordic Walking are recommended to patients with Type 2 Diabetes but their efficacy has not been demonstrated.

It is unknown whether one specific type of physical training program is more suitable than another, when comparing the physical effects as well as the ability to induce good compliance and change in lifestyle.

The aim of this randomized, controlled trial was to evaluate the effect of two different physical exercise programs lasting 4 months aiming at introducing long term life style changes in physical activity with a follow-up period of 8 months in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes for more than one year,
* HbA1c in the range of 7-10 %,
* BMI > 25 kg/m2,
* Age 25-80 years
* Stable antidiabetic treatment for at least 3 month before inclusion.

Exclusion Criteria:

* Participants with symptomatic heart disease (NYHA 2-4)
* Ischemia in lower extremities,
* Myocardial infarction within the previous 3 months
* Lung disease

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2005-02; Primary Completion 2006-10 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Glycated hemoglobin (HbA1c). | Baseline, after 4 months, after 1 year

SECONDARY OUTCOMES:
Adherence, Anthropometry,Blood pressure, Lipid profile, VO2max and quality of life. | Baseline, after 4 months, after 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bibi Gram, Ph.d student, Principal Investigator — University of Southern Denmark; Jeppe Gram, MD, Ph.d., Study Chair — Hospital of Southwest Denamark
Locations (1):
- Department of Endocrinology, Hospital of Southwest Denmark, Esbjerg, Region Syddanmark, Denmark